CLINICAL TRIAL: NCT03090659
Title: A Clinical Study of Legend Biotech BCMA-chimeric Antigen Receptor Technology in Treating Relapsed/Refractory (R/R) Multiple Myeloma Patients
Brief Title: LCAR-B38M Cells in Treating Relapsed/Refractory (R/R) Multiple Myeloma
Acronym: LEGEND-2
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanjing Legend Biotech Co. (Industry)
Collaborators: Second Affiliated Hospital of Xi'an Jiaotong University (Other); Ruijin Hospital (Other); Jiangsu Provincial People's Hospital (Other); Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCAR-B38M
Record Dates: First submitted 2017-03-07; First posted 2017-03-27 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Refractory or Relapsed Multiple Myeloma
Keywords: multiple myeloma; BCMA; CAR-T
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LCAR-B38M treatment group (Experimental): r/r multiple myeloma patients be treated with a split doses of LCAR-B38M cells. Total dose of 0.5-5 millions /kg cells will be administered at day 0, day 2 and day 6 by split dose (20%, 30% and 50% respectively).
  Interventions: Biological: LCAR-B38M CAR-T cell injection

INTERVENTIONS:
Biological: LCAR-B38M CAR-T cell injection

SUMMARY:
This is a single arm, open-label, multi-center, phase 1/2 study, to determine the safety and efficacy of LCAR-B38M CAR-T cells in treating patients diagnosed with refractory/relapsed multiple myeloma (r/r MM).

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a usually incurable malignancy of plasma cells. Current therapies for multiple myeloma often cause remissions, but nearly all patients eventually relapse and die, an clear unmet clinical needs. As early as mid-2014, the investigators have started to develop a series of proprietary CAR-T products to target B cell maturation antigen (BCMA), a cell surface molecule which the investigator believes to be a desirable target antigen for multiple myeloma. All pre-clinical data and CMC data for LCAR-B38M CAR-T cell technology has been established by mid-2015 and a phase I proof-of-concept clinical trial has been planned since then.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed prior diagnosis of active multiple myeloma as defined by the updated IMWG criteria.
* Patients with refractory multiple myeloma. Clear BCMA expression must be detected on malignant plasma cells from either bone marrow or a plasmacytoma by flow cytometry or immunohistochemistry.
* Refractory disease：1) At least 3 prior regimens, which must at least have contained bortezomi. or 2) other circumstances identified by clinical doctors.
* Relapse criteria in NCCN clinical practice guidelines in Oncology: Multiple Myeloma (2016.V2)

Exclusion Criteria:

* Women of child-bearing potential or who are pregnant or breastfeeding.
* Have any active and uncontrolled infection: hepatitis B, hepatitis C, HIV, or other fatal viral and bacterial infection.
* Systemic corticosteroid steroid therapy of greater than 5 mg/day of prednisone or equivalent dose of another corticosteroid are not allowed within 2 weeks prior to either the required leukapheresis or the initiation of the conditioning chemotherapy regimen.
* Patients with any uncontrolled intercurrent illness or serious uncontrolled medical disorder.
* Patients with CNS metastases or symptomatic CNS involvement (including cranial neuropathies or mass lesions and spinal cord compression).
* History of allogeneic stem cell transplantation. Have active acute or chronic graft-versus-host-disease (GVHD), or require immunosuppressant medications for GVHD, within 6 months of enrollment.
* Patients with active autoimmune skin diseases such as psoriasis or other active autoimmune diseases such as rheumatoid arthritis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-10-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment related adverse events as assessed by CTCAE v4.0 | Day 1-30 days after injection
  >= Grade 1 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment

SECONDARY OUTCOMES:
Anti-myeloma responses to LCAR-B38M cell treatment | Day 1-36 months after three split doses
  by measuring the changes of aberrant immunoglobulin in serum
Anti-myeloma responses to LCAR-B38M cell treatment | Day 1-36 months after three split doses
  multiple myeloma cells in bone marrow.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu J, Wang BY, Yu SH, Chen SJ, Yang SS, Liu R, Chen LJ, Hou J, Chen Z, Zhao WH, He AL, Mi JQ, Chen SJ. Long-term remission and survival in patients with relapsed or refractory multiple myeloma after treatment with LCAR-B38M CAR T cells: 5-year follow-up of the LEGEND-2 trial. J Hematol Oncol. 2024 Apr 24;17(1):23. doi: 10.1186/s13045-024-01530-z. PMID 38659046
- [Derived] Palmer S, Lin Y, Martin TG, Jagannath S, Jakubowiak A, Usmani SZ, Buyukkaramikli N, Phelps H, Slowik R, Pan F, Valluri S, Pacaud L, Jackson G. Extrapolation of Survival Data Using a Bayesian Approach: A Case Study Leveraging External Data from Cilta-Cel Therapy in Multiple Myeloma. Oncol Ther. 2023 Sep;11(3):313-326. doi: 10.1007/s40487-023-00230-x. Epub 2023 Jun 4. PMID 37270762
- [Derived] Zhao WH, Wang BY, Chen LJ, Fu WJ, Xu J, Liu J, Jin SW, Chen YX, Cao XM, Yang Y, Zhang YL, Wang FX, Zhang PY, Lei B, Gu LF, Wang JL, Zhang H, Bai J, Xu Y, Zhu H, Du J, Jiang H, Fan XH, Li JY, Hou J, Chen Z, Zhang WG, Mi JQ, Chen SJ, He AL. Four-year follow-up of LCAR-B38M in relapsed or refractory multiple myeloma: a phase 1, single-arm, open-label, multicenter study in China (LEGEND-2). J Hematol Oncol. 2022 Jul 6;15(1):86. doi: 10.1186/s13045-022-01301-8. PMID 35794616
- [Derived] Zhao WH, Liu J, Wang BY, Chen YX, Cao XM, Yang Y, Zhang YL, Wang FX, Zhang PY, Lei B, Gu LF, Wang JL, Yang N, Zhang R, Zhang H, Shen Y, Bai J, Xu Y, Wang XG, Zhang RL, Wei LL, Li ZF, Li ZZ, Geng Y, He Q, Zhuang QC, Fan XH, He AL, Zhang WG. A phase 1, open-label study of LCAR-B38M, a chimeric antigen receptor T cell therapy directed against B cell maturation antigen, in patients with relapsed or refractory multiple myeloma. J Hematol Oncol. 2018 Dec 20;11(1):141. doi: 10.1186/s13045-018-0681-6. PMID 30572922